CLINICAL TRIAL: NCT02166437
Title: Clinical Results of Bisphosphonate and Denosumab Therapy Following Teriparatide Therapy for Japanese, Prospective Study
Brief Title: Clinical Results of Bisphosphonate and Denosumab Therapy Following Teriparatide Therapy for Japanese
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tomidahama Hospital (Other)
Responsible Party: Principal Investigator, Toshihiko Kono, Head of Hospital, Tomidahama Hospital
Other Study IDs: IRB TH No 6-3
Record Dates: First submitted 2014-06-15; First posted 2014-06-18 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Osteoporosis
Keywords: osteoporosis; BMD; teriparatide; bisphosphonate; denosmab
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Alendronate: Patients treated with alendronate
- Minodronate: Patients treated with minodronate
- Denosmab: Patients treated with denosmab

SUMMARY:
In this study, the investigators would like to analyze the bone mineral density (BMD) , bone turnover makers, and fracture prevention effects of bisphosphonate and denosumab randomly divided following daily teriparatide in Japanese patients under clinical practice. The participants are treated in the investigators hospital, who are under severe osteoporotic condition.

DETAILED DESCRIPTION:
Registry criteria: Patients treated in the investigators hospital using teriparatide. Enrolled patients are severe osteoporosis; more than two previous osteoporotic fractures, low BMD (< young adult mean 65%).

Interventions: blood analyses and dual-energy X-ray absorptiometry (DXA) every 4 months Informed consent: Written informed consent will be obtained. Sample size: Five-hundreds participants

ELIGIBILITY:
Inclusion Criteria:

* severe osteoporotic patients

Exclusion Criteria:

* cancer, hypercalcemia, etc (i.e. patients who could not use bisphosphonate, denosmab, teriparatide)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: tion Osteoporotic patients who admit to our hospital
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Clinical results of bisphosphonate vs. denosmab following daily teriparatide treatment | Up to 36 months
  The investigators plan to analyze 500 patients who treated with bisphosphonate or denosmab following daily teriparatide treatment.
  We investigate changes in BMD and bone turnover markers.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Niimi, MD, PhD, Study Director — Tomidahama Hospital
Locations (1):
- Tomidahama Hospital, Yokkaichi, Mie-ken, Japan